CLINICAL TRIAL: NCT00421824
Title: Phase II Randomized Trial of Neoadjuvant Chemotherapeutic Treatment (XELOX) Followed by Chemoradiotherapy (XELOX/RT) and Surgery Versus Chemoradiotherapy Followed by Surgery and Chemotherapy in Patients With High Risk Rectal Cancer
Brief Title: Study of Neoadjuvant Chemotherapeutic Treatment (XELOX) Followed by Chemoradiotherapy (XELOX/RT) and Surgery Versus Chemoradiotherapy Followed by Surgery and Chemotherapy in Patients With High Risk Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0098; EudraCT # : 2005-005149-20
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy

ARMS (2):
- A (Experimental)
  Interventions: Drug: Oxaliplatin, capecitabine
- B (Experimental)
  Interventions: Drug: Oxaliplatin, capecitabine

INTERVENTIONS:
Drug: Oxaliplatin, capecitabine — OXA 130 D1 + Capecitabine 2000 / day D1-D14 for 4 cycles. After 10 weeks of rest, XELOX-RT regimen x 5 weeks followed by surgery
  Other Names: Radiotherapy
  Arms: A
Drug: Oxaliplatin, capecitabine — XELOX-RT x 5 weeks followed by surgery and 4 cycles of adjuvant XELOX with the same scheme as arm A.
  Other Names: Radiotherapy
  Arms: B

SUMMARY:
Primary:

* To assess complete pathological response rate of both strategies.

Secondary:

* Safety profile
* To assess downstaging rate of both strategies.
* To compare relative dose intensity of oxaliplatin and capecitabine of both strategies
* To compare time to progression and overall survival of both strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal adenocarcinoma.
* Operable tumour, confirmed by magnetic resonance of high resolution and / or endorectal echography, or,
* Rectal tumour at distal third, or
* Tumours spread more than 5 mm in perirectal fat
* Functional state ECOG ≤ 2.
* Good hematological, hepatic and renal function

Exclusion Criteria:

* Previous pelvis radiotherapy.
* Previous antitumoural chemotherapy
* Pregnant or breastfeeding women.
* Childbearing women with a positive pregnancy test result at baseline. Menopausal women should not have the period for the last 12 months.
* History of any other neoplastic illness within the last 5 years, except for already resolved small cell skin cancer or cervix cancer.
* Clinically significant cardiovascular disease
* Confirmed peripheral neuropathy.
* Gastrointestinal disorders or bad absorption syndrome or non-capable to take oral medication.
* Blood disorders.
* Intercurrent non-controlled or severe infections.
* Patients who have undergone major surgery, open biopsies or with significant trauma lesions within the previous 28 days.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Response rate | from the signature of Informed Consent up to the end of the study

SECONDARY OUTCOMES:
Relative dose intensity | from the signature of Informed Consent up to end of the study
Disease free survival | from the signature of Informed Consent up to end of the study
Overall survival | from the signature of Informed Consent up to end of the study

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Taboada, Dr., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Barcelona, Spain